CLINICAL TRIAL: NCT00254449
Title: A Randomized, Controlled, Open-Label Study to Investigate the Effect of NGX-4010 on Epidermal Nerve Fiber Density and Sensory Function in Healthy Volunteers
Brief Title: Effect of NGX-4010 on ENFD and Sensory Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeurogesX (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C115
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2007-09

CONDITIONS: Human Volunteers
MeSH Terms: interventions — Capsaicin

INTERVENTIONS:
Drug: NGX-4010

SUMMARY:
The purpose of this study is to evaluate epidermal nerve fiber (ENF) regeneration and normalization of peripheral sensory nerve function over time in normal healthy volunteers following a 60 minute application of Capsaicin Dermal Patch (NGX 4010; capsaicin 640 mcg/cm2) as compared to comparable untreated skin areas (control).The objectives of this study are: 1) To assess the difference between patch-treated and comparable untreated skin areas (control) in ENFD as quantified by PGP 9.5 immunohistochemical staining of skin biopsy samples obtained at 1, 12 and 24 weeks following a 60 minute application; 2) To assess the difference between patch-treated and comparable untreated skin areas (control) for thermal detection thresholds as assessed by QST at 1, 12 and 24 weeks following a 60 minute application; and, 3) To assess the difference between patch-treated and comparable untreated skin areas (control) in mechanical (sharp pain) sensation and tactile threshold at 1, 12 and 24 weeks following a 60 minute application.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, single center, phase 1 study in normal healthy volunteers. Each subject will have a 60 minute exposure to two 5.0 × 5.5 cm NGX-4010 patches. In addition, two 5.0 × 5.5 cm comparable untreated control skin areas will be identified and evaluated. At baseline and prior to skin punch biopsy at Weeks 1 (± 1 day), 12 (± 3 days) and 24 (± 7 days), QST of patch-treated and untreated control skin areas will be performed and evaluated. QST for cooling detection threshold and heat-pain threshold, and assessment of mechanical (sharp pain) sensation and tactile threshold will be performed at each of the two patch-treated and two untreated control skin areas. Serial skin punch biopsies of patch-treated and untreated control skin areas will be obtained and evaluated at Weeks 1 (± 1 day), 12 (± 3 days), and 24 (± 7 days). Skin at the patch-treated and untreated control skin areas will be anesthetized with subcutaneous 1% lidocaine, and then three millimeter (mm) skin biopsies will be obtained with a sterile punch tool from each of the designated areas. Biopsy specimens will be fixed overnight, then cryoprotected in a phosphate buffered solution until processed. Thick sections will be cut and immunostained for localization and quantification of nerve fibers in the epidermis and visualization of the subepidermal plexus using antibodies to PGP 9.5. Antibodies to type IV collagen will be used to identify the basement membrane and superficial blood vessels in the biopsy microsections. Vital signs and adverse events (AEs) will be collected at each visit. Clinical laboratory tests will be performed at the Screening Visit and at the Termination Visit (Week 24).

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years of age.
* Male and female subjects. (Half of the subjects enrolled must be male.)
* Be in good health.
* Have intact, unscarred skin over the thighs.
* Agree not to use topically-applied products containing nonsteroidal antiinflammatory drugs, menthol, methyl salicylate, local anesthetics, steroids or capsaicin anywhere on the thighs for the duration of the study.
* Female subjects must not be breast-feeding and must have a negative serum beta human chorionic gonadotropin (hCG) pregnancy test performed within 7 days prior to the Study Patch Application Visit (Day 0).
* All subjects must be willing to use effective methods of birth control and/or refrain from participating in a conception process during the study and for 30 days following experimental drug exposure.
* Willing and able to comply with protocol requirements for the duration of study participation. Requirements include but are not limited to attending all study visits and refraining from extensive travel during study participation.
* Subjects must sign an informed consent form for this study approved by the Investigator's Institutional Review Board (IRB).

Exclusion Criteria:

* Any dermatological condition(s) that in the judgment of the Principal Investigator has the potential to disrupt skin integrity or alter sensory function on the thighs.
* Any skin infection, skin irritation (e.g., poison oak), trauma or burn (including sunburn) on the thighs within 30 days preceding the Study Patch Application Visit (Day 0).
* Any medical history of painful conditions, surgery, or injury involving or affecting the thighs, including but not limited to prior orthopedic surgery, lumbosacral disc disease, sciatica, and hip or femur fracture.
* Any medical history of known or suspected body system abnormalities, including but not limited to diabetes, hypothyroidism, asthma or any form of peripheral or central nervous system disease.
* Use of any systemic medications that interact with the peripheral nervous system, including beta adrenergic blockers, alpha adrenergic blockers, anticonvulsant drugs, antidepressant drugs or opioids within 30 days prior to the Study Patch Application Visit (Day 0).
* Use of any topically-applied product including prescription or over the-counter (OTC) analgesic creams/lotions/patches, nonsteroidal antiinflammatory drugs, local anesthetics, steroids or capsaicin on the thighs within 30 days preceding the Study Patch Application Visit (Day 0).
* Currently taking any prescription medication except for oral, transdermal or injected contraceptives.
* Requirement for ongoing or periodic pain medication for any chronic or recurrent medical condition.
* Participation in another drug research study within 30 days preceding the Study Patch Application Visit (Day 0).
* Diagnosis of human immunodeficiency virus (HIV) infection, according to medical history and/or self-report.
* History or current substance abuse including alcoholism/alcohol abuse, as judged by the investigator.
* Positive test result on the urine drug screen for opioids, cannabis, phencyclidine (PCP), cocaine and amphetamines performed at the Screening Visit.
* History of hypersensitivity to capsaicin (i.e., chili peppers or OTC capsaicin products), local anesthetics including lidocaine or adhesives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2005-11; Study Completion 2006-05

PRIMARY OUTCOMES:
Mean ENFD in the patch-treated and comparable untreated skin areas (control) at 1, 12 and 24 weeks after exposure.
Mean just noticeable difference (JND) values for thermal perception QST in the patch-treated and comparable untreated skin areas (control) at 1, 12 and 24 weeks after exposure.
Mean difference in mechanical (sharp pain) sensation and tactile threshold between patch-treated and comparable untreated skin areas (control) at 1, 12 and 24 weeks after exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Tobias, MD, Study Director — NeurogesX; William R. Kennedy, MD, Principal Investigator — University of Minnesota
Locations (1):
- NeurogesX Investigational Site, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Kennedy WR, Vanhove GF, Lu SP, Tobias J, Bley KR, Walk D, Wendelschafer-Crabb G, Simone DA, Selim MM. A randomized, controlled, open-label study of the long-term effects of NGX-4010, a high-concentration capsaicin patch, on epidermal nerve fiber density and sensory function in healthy volunteers. J Pain. 2010 Jun;11(6):579-87. doi: 10.1016/j.jpain.2009.09.019. Epub 2010 Apr 18. PMID 20400377